CLINICAL TRIAL: NCT03521518
Title: Neuropsychometric Testing With Conner's Continual Performance Test -3 in Normal Pressure Hydrocephalus
Brief Title: CPT-3 in Normal Pressure Hydrocephalus
Status: Terminated | Type: Observational
Why Stopped: Inadequate enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Eaton, Principle Investigator, Vanderbilt University Medical Center
Other Study IDs: VR52393
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Normal Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Conner's Continuous Performance Test-3 — CPT-3 allows quantitative assessment of visuospatial, attention and reaction time in patients being evaluated for Normal Pressure Hydrocephalus undergoing a CSF tap test.

SUMMARY:
The study will collect prospective cohort data of individuals that are undergoing routine clinical care for suspected idiopathic Normal Pressure Hydrocephalus (NPH). The administration of the Conner's Continual Performance Test - version 3 (CPT-3), an automated 14-minute computerized measure of reaction-time and sustained attention, will be added to the current neurocognitive screen being used (i.e., the Montreal Cognitive Assessment, MoCA) along with gait assessment. Patients will undergo pre-tap testing on the morning of their large volume Lumbar Puncture (CSF-TT). These patients will receive post-tap CPT-3 and MoCA testing one-to-three hours post-tap, and again at 2-3 days post-CSF-TT, during the follow-up appointment in clinic.

The standard NPH quantitative assessment methods of MoCA and gait evaluation will continue to be collected. For those patients that ultimately undergo ventricular shunt placement, the CPT-3 will be administered at their post-operative follow-up appointment (~3 months post-operation). The results of CPT-3 will not factor into consideration for shunt candidacy.

DETAILED DESCRIPTION:
Normal pressure hydrocephalus (NPH) is a syndrome involving the clinical triad of gait disturbance, urinary incontinence, and cognitive dysfunction, in the context of ventricular enlargement out of proportion to parenchymal atrophy with normal intracranial pressure.

In the 1980's, a protocol for quantitative measurement of symptom response to large volume CSF tap (40-50ml) was developed, as a method for evaluating suitability for undergoing ventricular shunting surgery. A 2016 systematic review of the literature noted heterogeneous findings within the eight prospective cohort studies that were included in analysis, but concluded that there appeared to be support for the CSF-TT as a rule-in screen for response to shunt placement.

Unfortunately, no extant literature has analyzed the independent predictive power of a clinically significant reaction time improvement in response to CSF-TT (widely defined across the literature as 5% improvement) to subsequent response to ventricular shunting. This frustrates an a priori power analysis. However, a rough estimate was calculated based on data presented within one of the aforementioned reviewed studies that identified an improvement in reaction time in response to CSF-TT, as well as an improvement in reaction time to subsequent shunting.

The authors reported that 17 of 68 (25%) of the patients were labeled as positive-responders to CSF-TT, defined as meeting at least 2 of the following criteria: 1) 5% improvement in reaction time, 2) 5% improvement in gait (time or steps), 3) 25% improvement on visuospatial recall task, 4) 25% improvement on visuospatial recognition task. Of those 17 positive responders, 16 (94%) met the same positive-response criteria, post-shunting. If we use a 50% response rate as a proportion null hypothesis, this gives us a z-statistic = 3.63, or f2 = 3.71. G*Power analysis, for a 4-predictor regression (i.e., the aforementioned indicators used), estimates a necessary sample size of 16. The primary limitation of this approach is that it is unclear which of the 2+ positive response criteria were met. However, review of the pre- versus post-shunting data suggests reaction time was significantly improved (p<0.001; Cohen's d = 0.399), suggesting it is reasonable to infer the domain was favorably impacted by the temporary effects of a CSF-TT.

Patients will undergo pre-tap testing on the morning of their CSF-TT. The administration of the Conners Continual Performance Test - version 3 (CPT-3), an automated 14-minute computerized measure of reaction-time and sustained attention, will be added to the current neurocognitive screen being used (i.e., the Montreal Cognitive Assessment, MoCA). The current CSF-TT protocol's quantitative methods for measuring urinary incontinence and gait will continue to be collected. These patients will receive post-tap CPT-3 and MoCA testing one-to-three hours post-tap, and again at 2-3 days post-CSF-TT, during the follow-up appointment with Neurosurgery. For those that undergo ventricular shunt placement, the CPT-3 will be administered at their post-operative follow-up appointment (~3 months post-operation).

ELIGIBILITY:
Inclusion Criteria:

* patients being referred for CSF tap test as part of routine clinical assessment of idiopathic Normal Pressure Hydrocephalus by their medical provider
* adults older than 18 years old

Exclusion Criteria:

* premorbid neurodegenerative disease (e.g. Alzheimer's Disease, Frontotemproal Dementia, Parkinson's Disease)
* serious acquired brain injury such as moderate to severe traumatic brain injury, large ischemic strokes
* seizure disorders
* serious neuropsychiatric disease (e.g. schizophrenia, bipolar disorder, major depressive disorder, active alcohol or drug abuse)
* untreated vitamin deficiencies (B12, Wernicke-Korsakoff Syndrome)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with a clinical concern for Normal Pressure Hydrocephalus. They will be adults with cognitive impairment with at least one of the following: ventriculomegaly out of proportion to sulcal atrophy on imaging, urinary incontinence and problems with gait (magnetic gait or "apraxic gait").
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Attention and Responsiveness | 1-3 hours after lumbar puncture, 2-3 days after lumbar puncture
  5% Improvement in T-scores of patients after large volume lumbar puncture

SECONDARY OUTCOMES:
Attention and Responsiveness after Ventricular Peritoneal Shunt Placement | Approximately 3-6 months after VPS placement
  Patients that have VPS placed will be reassessed and again will be looking for improvement in T-scores.

CONTACTS AND LOCATIONS:
Overall Officials: James E Eaton, MD, Principal Investigator — Resident Physician
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hakim S, Adams RD. The special clinical problem of symptomatic hydrocephalus with normal cerebrospinal fluid pressure. Observations on cerebrospinal fluid hydrodynamics. J Neurol Sci. 1965 Jul-Aug;2(4):307-27. doi: 10.1016/0022-510x(65)90016-x. No abstract available. PMID 5889177
- [Background] Wikkelso C, Andersson H, Blomstrand C, Lindqvist G. The clinical effect of lumbar puncture in normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 1982 Jan;45(1):64-9. doi: 10.1136/jnnp.45.1.64. PMID 7062072
- [Background] Mihalj M, Dolic K, Kolic K, Ledenko V. CSF tap test - Obsolete or appropriate test for predicting shunt responsiveness? A systemic review. J Neurol Sci. 2016 Mar 15;362:78-84. doi: 10.1016/j.jns.2016.01.028. Epub 2016 Jan 22. PMID 26944123
- [Background] Kahlon B, Sundbarg G, Rehncrona S. Comparison between the lumbar infusion and CSF tap tests to predict outcome after shunt surgery in suspected normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):721-6. doi: 10.1136/jnnp.73.6.721. PMID 12438477